CLINICAL TRIAL: NCT04402710
Title: Examining the Feasibility and Acceptability of a Self-compassion Intervention on Physical Activity Behaviour Among People With Prediabetes
Brief Title: Is Teaching People to be Self-compassionate Feasible and Acceptable for People Who Are Pre-diabetic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E2020:006
Record Dates: First submitted 2020-04-09; First posted 2020-05-27 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2020-03

CONDITIONS: PreDiabetes
Keywords: self-compassion; physical activity; self-regulation; randomized controlled trial; emotions; feasibility; acceptability
MeSH Terms: conditions — Prediabetic State; Motor Activity; Self-Control | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either a control group or the intervention group. Both sessions will run concurrently.
Who Masked: Participant, Outcomes Assessor
Masking Description: The research assistant who is in charge of conducting the statistical analyses will not be involved in the randomization process or running the intervention or control groups.
  Research assistants who will be conducting in-person eligibility and/or follow-up visits (e.g. handing out accelerometers) will be blinded to participant group assignment.
  Participants will also be blinded to which group they are randomized into. The investigators will present the study as examining different education interventions to increase physical activity and will not let the participants know whether they are in the intervention or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Session 1: Participants will meet individually with a research assistant to discuss their type 2 risk and discuss benefits of engaging in 150 minutes of moderate-to-vigorous physical activity per week. Ideal Care will involve: Session 2: Introductions and Goal setting/planning. Session 3: Action-Coping Planning and Monitoring Physical Activity Session 4: Goal re-visitation and adjustment and building self-efficacy. Session 5: Physical Activity Enjoyment and Barriers/Solutions. Session 6: Relapse prevention and commitment to exercise. The last 30 minutes of sessions 2-6, control participants will receive 30-minutes of non-self-compassion or physical activity related health education (i.e., sleep, screen time, antibiotic use, oral health, osteoporosis and vitamin D).
  Interventions: Behavioral: Control Group
- Intervention Group (Experimental): Session 1: Participants will meet individually with a research assistant to discuss their type 2 risk and discuss benefits of engaging in 150 minutes of moderate-to-vigorous physical activity per week. First 30 minutes of each subsequent session will be ideal care (as described above in the control group). Last 30 minutes of sessions 2-6, self-compassion condition participants will learn to apply self-compassion to their prediabetes experience and physical activity. Session 2: Learn about fear of self-compassion and the benefits of self-compassion. Session 3: Yin and Yang of self-compassion. Session 4: Mindfulness. Session 5: Dealing with difficult emotions, loving Kindness and Self-Compassionate motivation. Session 6: Living deeply, self-appreciation and stages of progress.
  Interventions: Behavioral: Self-compassion

INTERVENTIONS:
Behavioral: Self-compassion — Six week behavioural change program plus a self-compassion intervention aimed to increase physical activity among individuals with prediabetes
  Arms: Intervention Group
Behavioral: Control Group — Six week behavioural change program aimed to increase physical activity plus information on general health topics.
  Arms: Control Group

SUMMARY:
The investigators plan to examine the feasibility and acceptability of an online, two arm intervention ([self-compassion intervention + ideal care] versus [health information + ideal care]) designed to increase physical activity among individuals at risk of type two diabetes. The aim of the self-compassion intervention is to teach people at risk of type two diabetes how to use self-compassion (orientation to care for oneself during difficult situations) in order to help them self-manage and increase their physical activity. In a group, online format people at risk for type 2 diabetes will learn about their type 2 diabetes risk and strategies to increase their physical activity, which represents the recommended information that people at risk for type two diabetes should receive (i.e. ideal care). In addition to this, some participants, but not all, will be taught to be self-compassionate in relation to their type two diabetes risk and their efforts to increase their physical activity (i.e. intervention group). The other participants (i.e. control group) will instead receive general health information in addition to ideal care. Feasibility outcomes will be assessed using Thabane and colleagues (2010) model including the study's process, resources, management and scientific outcomes. In addition, qualitative exit-interviews with participants and research personnel will be conducted to assess the acceptability and feasibility of the intervention. Lastly, investigators will explore whether the intervention leads to changes from pre- to post-intervention in the secondary outcomes. This study is important as it will help inform and ensure the larger efficacy trial is of high quality.

DETAILED DESCRIPTION:
The primary research objective of this study is to test the feasibility and acceptability of an online, two arm ([self-compassion intervention + ideal care] versus [health information + ideal care]) intervention designed to increase physical activity among individuals at risk for type 2 diabetes.

Primary research question: Is an online, two-arm intervention ([self-compassion intervention + ideal care] versus [health information + ideal care]) focused on increasing physical activity levels among individuals at risk of type two diabetes feasible using Thabane and colleagues model of feasibility (2010)?

Secondary research question: Is an online, two-arm intervention ([self-compassion intervention + ideal care] versus [health information + ideal care]) focused on increasing physical activity levels among individuals at risk of type two diabetes acceptable to both participants and research personnel?

The secondary research objective is to explore whether an online, two-arm intervention ([self-compassion intervention + ideal care] versus [health information + ideal care]) focused on increasing physical activity levels among individuals at risk of type two diabetes leads to changes from pre- to post-intervention in self-compassion, physical activity levels, nutrition, self-regulatory skill use, experience of exercise barriers, personal growth initiative, negative affect, and engagement in other health behaviours (e.g. stress management).

This pilot and feasibility study is a single centre, randomized, active controlled, six week intervention with baseline and follow-up assessment at intervention-end, 6- and 12-weeks post-intervention. It follows a quantitative-dominant, mixed-methods design. They will supplement this trial with interviews after follow-up testing with participants and study personnel. These interviews will provide feasibility and acceptability information.

ELIGIBILITY:
Inclusion Criteria:

* Medium to high type 2 diabetes risk (assessed with the CANRISK tool)
* Age 40 - 74
* No current medical treatment for type 2 diabetes
* Safe to engage in physical activity
* No non-study self-reported current type 2 diabetes/behaviour change education that may interfere with the intervention
* Available for all sessions and testing
* Insufficient physical activity relative to guidelines of 150 minutes of moderate to vigorous physical activity per week.
* Below the mean on the self-compassion scale

Exclusion Criteria:

* Be under 40 years old, or over the age of 74
* Have a medical condition which would not allow them to participate safely in physical activity
* Already are part of a different behavioural change/ type 2 diabetes education group
* Already engage in over 150 minutes of moderate to vigorous physical activity per week
* Already have high levels of self-compassion (over the mean)
* Could not commit to the intervention/control sessions

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | During the recruitment phase of the study
  Number of participants screened/showed interest in partaking in the study during the recruitment period and how many of these individuals get successfully recruited into the study.
Most successful Recruitment Strategy | During the recruitment phase of the study
  Participants will be asked to state how they heard about the study
Retention Rates | Week 1 (baseline) to Week 18 (follow-up)
  The number of people who begin the study relative to the number of people who drop out at any point during the study.
Compliance | Week 1 (baseline) to Week 18 (follow-up)
  This will consist of online class attendance and through participant responses using a text messaging system (e.g. responding 'yes' or 'no' to whether they completed their at home practice), and will be determined by the number of individuals who wear their accelerometer for the recommended 4 days, 10 hours per day.
Instructor Fidelity | Week 1 (baseline) to Week 6 (end of intervention)
  How well facilitators conduct class sessions and activities compared to the set protocol. This will be determined by a checklist with a protocol for each session where facilitators will identify what components they did/did not complete and whether they followed the session protocol accordingly. With participant approval, facilitators will video record 15% of all sessions and the principal investigator will assess the adherence to the planned intervention, presentation skills, and will assess the adherence to the planned intervention, presentation skills, and will rate communication skills. The principal investigator will rate each component on a 5-point Likert scale.
Capacity | Week 1 (baseline) to Week 18 (follow-up)
  This will be determined by evaluating whether the number of hours it takes study personnel to complete study tasks stays under the total cost that was budgeted for personnel hours for this study.
Process Time | During the recruitment phase of the study
  How much time it takes to send out the initial eligibility email questionnaire, determine the participant's eligibility, and contact the eligible participant for the next steps of the study.
Study Personnel Challenges and Insights | 6 weeks (end of intervention)
  Through a semi-structured exit-interview study personnel will be asked whether they encountered any challenges throughout the study or have any reccomendations.
Participant safety will be assessed by asking participants to explain their thoughts and feelings about whether the study impacted their physical and psychological safety through a semi-structured exit interview. | 6-weeks (end of intervention)
  To determine whether participants felt safe while participating in this study, they will be asked to explain their thoughts and feelings through a semi-structured exit-interview. A sample question is, "Did you feel safe physically and psychologically during each session"
Acceptability as assessed by semi-structured exit interviews with participants which will include questions related to their thoughts and feelings about the study and whether they believed the study was acceptable (e.g. content, timing). | 6 weeks (end of intervention)
  To assess participant satisfaction and their experience with the study, they will be asked a variety of questions to understand their thoughts and feelings during the semi-structured exit-interview. An example question participants will be asked is, "what components of the intervention did you like/dislike?"

SECONDARY OUTCOMES:
Change in Moderate to Vigorous Physical Activity from baseline to 6 weeks (intervention end) | baseline to 6 weeks (intervention end)
  Physical activity as measured by GT3X+ accelerometers (1952 - >9498 counts per min)
Change in self-report Moderate to Vigorous Physical Activity from baseline to 6 weeks (intervention end) | baseline to 6 weeks (intervention end)
  Physical activity as measured by GT3X+ accelerometers (1952 - >9498 counts per min)
Change in Self-Compassion from baseline to 6 weeks (intervention end) | baseline to 6 weeks
  Self-Compassion Scale (Neff, 2003); 6-point Likert scale ranging from a mean value of 1 (low self-compassion) to 5 (high self-compassion)
Change in Mild Physical Activity from baseline to 6 weeks (intervention end) | baseline to 6 weeks (intervention end)
  Measured by GT3X Accelerometers (100 - 1952 counts per min)
Change in Sporadic Physical Activity from baseline to 6 weeks (intervention end) | baseline to 6 weeks (intervention end)
  Measured by GT3X Accelerometers (bouts of moderate to vigorous physical activity less than 10 minutes with no drop in intensity)
Change in Negative Affect Related to Diabetes Risk from baseline to 6 weeks (intervention end) | baseline to 6-weeks (intervention end)
  Negative Affect Scale (Leary, Tate, Adams, Allen, & Hancock, 2007); 7-point Likert scale ranging from 1 (not at all) to 7 (Extremely); Scale Range: 20 (low Negative Affect) - 140 (high Negative Affect)
Change in Negative Affect Related to Low Physical Activity Levels from baseline to 6 weeks (intervention end) | 6-weeks (intervention end)
  Negative Affect Scale (Leary, Tate, Adams, Allen, & Hancock, 2007); 7-point Likert scale ranging from 1 (not at all) to 7 (Extremely); Scale Range: 20 (low Negative Affect) - 140 (high Negative Affect)
Change in Health Promoting Behaviors from baseline to 6 weeks (intervention end) | baseline to 6 weeks (intervention end)
  Health-Promoting Lifestyle Profile II (Walker, Sechrist, & Pender, 1995); 4-point Likert scale ranging from 1 (never) to 4 (routinely); Scale range: 52 (low engagement in health behaviours) to 208 (high engagement in health behaviours)
Change in Fear of Self-Compassion from baseline to 6 weeks (intervention end) | baseline week 1
  Fear of Self-compassion Scale (Gilbert et al., 2011); 5-point Likert scale ranging from 0 (not fearful) - 60 (very fearful)
Change in Exercise barriers from baseline to 6 weeks (intervention end) | baseline to 6 weeks (intervention end).
  Exercise Barrier Scale (Sechrist et al., 1987). 4-point Likert scale ranging from 1 (strongly agree) to 4 (strongly disagree); 14 items; participants are asked to indicate the degree to which they have different barriers to exercise. Higher scores indicate less exercise barriers. Overall score ranges from 14 to 56.
Change in Cognitive Emotion Regulation strategies from baseline to 6 weeks (intervention end) | baseline to 6 weeks (intervention end)
  Cognitive Emotion Regulation Questionnaire (Garnefski et al. 2001). 5-point Likert scale ranging from 1 (almost never) to 5 (almost always); 36 items; Participants are asked the extent to which they make use of certain cognitive coping strategies. Nine different subscales: self-blame, other-blame, rumination, catastrophizing, putting into perspective, positive refocusing, positive reappraisal, acceptance, refocus on planning. Each subscale is totaled with higher scores indicating higher use of that cognitive emotional strategy. Scores for each subscale can range from 4 to 20.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Signore AK, Jung ME, Semenchuk B, Kullman SM, Tefft O, Webber S, Ferguson LJ, Kowalski K, Fortier M, McGavock J, Ahmed R, Orr M, Strachan S. A pilot and feasibility study of a randomized clinical trial testing a self-compassion intervention aimed to increase physical activity behaviour among people with prediabetes. Pilot Feasibility Stud. 2022 May 27;8(1):111. doi: 10.1186/s40814-022-01072-6. PMID 35624519